CLINICAL TRIAL: NCT00866827
Title: Airway Vascular Lesions
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 20969; Unfunded, Retrospective review
Record Dates: First submitted 2007-12-17; First posted 2009-03-23 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Hemangiomas; Venous Malformations; Lymphatic Malformations
Keywords: Airway; Hemangiomas; Venous Malformations; Lymphatic Malformations
MeSH Terms: conditions — Hemangioma; Lymphatic Abnormalities | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Other: Protocols for Treatment — Determine protocols for treatment of airway vascular malformation and to evaluate results from treatment of these lesions.

SUMMARY:
Controversy exists in the treatment of airway hemangiomas ranging from tracheotomy, various lasers, to open removal, none of which have proven to be a gold standard. Venous malformations of the airway are difficult to treat and also require laser therapy or open removal and often repeated treatments are required. Similarly airway lymphatic malformations can require multiple treatment modalities as well as multiple procedures and are infrequently eradicated when extensive. New uses for various lasers and differing treatment protocols are frequently developed. Review of the treatment modalities and efficacy of these methods is required. The goal of this research is to determine protocols for treatment of airway vascular malformation and to evaluate our results from treatment of these lesions.

ELIGIBILITY:
Inclusion Criteria:

* Airway Vascular Lesion

Exclusion Criteria:

* None at this time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in the ACH database that have been treated in the last ten years for airway vascular lesions.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2002-12; Primary Completion 2014-04-15 (Actual); Study Completion 2014-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gresham T Richter, M.D., Principal Investigator — UAMS, ACH, Central Arkansas Veterans Healthcare System; Jessica L Boswell, BS, CRS, Study Director — UAMS, ACH, Central Arkansas Veterans Healthcare System